CLINICAL TRIAL: NCT06196385
Title: Efficacy Of Intensive Cervical Traction On Depression, Insomnia, Quality of Life In Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moataz Mohamed Talaat El Semary, Assistant Professor of physical therapy for neurology and neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004910
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Traction; Depression; insomnia; Quality of life
MeSH Terms: conditions — Radiculopathy; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: post hoc test
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive Cervical Traction for cervical radiculopathy (Experimental): Using intensive cervical traction through mechanical computerized device
  Interventions: Device: intensive Cervical Traction
- intensive Cervical Traction for healthy matched group (Active Comparator): USING TRACTION FOR HEALTHY MATCHED AGE CONTROL GROUP
  Interventions: Device: intensive Cervical Traction

INTERVENTIONS:
Device: intensive Cervical Traction — A 30-minute cervical traction protocol, twice a day, for five consecutive days per week for 6 weeks. The main objective will be the evaluation of depression, insomnia, and quality of life. We evaluate at prior to the treatment and, at the end of the protocol, for depression, insomnia, and quality of life.

SUMMARY:
Cervical radiculopathy is a common and disabling condition involving local pain in the neck region and pain that radiates into the upper limb. Recent data suggest that cervical traction may effectively reduce disability and pain, with a dose-response relationship. The main aim of this study was therefore to evaluate the effect of an intensive cervical traction protocol for patients with cervical radiculopathy on depression, insomnia, and quality of life (1).

DETAILED DESCRIPTION:
The investigators will conduct a prospective open observational study of thirty-six patients referred by their neurosurgeons for symptoms suggestive of cervical radiculopathy. All patients undergo the same treatment: a 30-minute cervical traction protocol, twice a day, for five consecutive days per week for 6 weeks. The main objective will be the evaluation of depression, insomnia, and quality of life. The investigators will evaluate at prior to the treatment and, at the end of the protocol, for depression, insomnia, and quality of life. The primary outcomes will be hospital anxiety and depression scale (HADS) and Short Form 36 Health Survey (SF-36) before and after treatment with spinal traction. Thirty-five healthy controls, matched with patients for age and sex, completed the same questionnaires. Traction was added to patients' medications which were not enough to control patients' symptoms and did not change during traction.

Depressive and anxiety symptoms were assessed by an Arabic version of Hospital Anxiety and Depression scale. Health-related quality of life was assessed by applying the Arabic version of the Short-Form 36 Health Survey (SF-36) [ Insomnia severity index will be used to evaluate insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prolapsed cervical disc were diagnosed based on clinical examination and MRI cervical spine
* Patients showed only some improvement on medical treatment, NSAI drugs, muscle relaxants, and drugs for neuropathic pain, which will continue and will not change during spinal traction

Exclusion Criteria:

* In addition to non-consenting patients, patients with the following conditions will be excluded from the present study: ligamentous instability, osteomyelitis, diskitis, primary or metastatic spinal cord tumor, severe osteoporosis, myelopathy, fibromyalgia, or untreated hypertension.
* Patients currently treated for psychiatric disorders, or those who had past history of psychiatric disorders, will also excluded

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — ISLAMIC ISSUES MORE SPECIFIC FOR HOMOGENITY
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Hospital anxiety and depression scale (HADS) | before and after 6 WEEKS OF treatment with spinal traction
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire that has been found to be a reliable instrument for detecting states of anxiety and depression in the setting of hospital outpatient clinic. The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Short Form 36 Health Survey (SF-36) | before and after 6 WEEKS OF treatment with spinal traction
  Qualiveen short version 8 questions from 1 to 4 (worse if high score)
Insomnia severity index | before and after 6 WEEKS OF treatment with spinal traction
  Though developers point out that their chosen cutoff scores have not been validated, they offer a few guidelines for interpreting scale results: a total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "subthreshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
NO sharing to keep confidentiality

REFERENCES:
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Van't Veer A, Yano JM, Carroll FI, Cohen BM, Carlezon WA Jr. Corticotropin-releasing factor (CRF)-induced disruption of attention in rats is blocked by the kappa-opioid receptor antagonist JDTic. Neuropsychopharmacology. 2012 Dec;37(13):2809-16. doi: 10.1038/npp.2012.151. Epub 2012 Sep 5. PMID 22948977
- [Background] Oktay EA, Ersahan S, Gokyay S. Effect of intracanal medicaments used in endodontic regeneration on the push-out bond strength of a calcium-phosphate-silicate-based cement to dentin. Pak J Med Sci. 2018 Mar-Apr;34(2):310-315. doi: 10.12669/pjms.342.14630. PMID 29805399